CLINICAL TRIAL: NCT00499343
Title: A Randomized Study Comparing Chemotherapy Followed by G-CSF Alone Versus G-CSF Plus GM-CSF for Mobilization of Peripheral Blood Stem Cells in Patients With Non-Hodgkin's Lymphomas
Brief Title: G-CSF Versus G-CSF Plus GM-CSF for Stem Cell Mobilization in NHL Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0242
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Results first posted 2009-07-07 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Lymphoma; Etoposide; G-CSF; GM-CSF; Isophosphamide; Rituximab; Ifosfamide; Sargramostim; Leukine; Filgrastim; Neupogen; Apheresis; Stem Cell Collection
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Etoposide; Granulocyte Colony-Stimulating Factor; Filgrastim; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Ifosfamide; Rituximab; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab + Ifosfamide + Etoposide + 2 Growth Factors (Experimental): Growth Factors = granulocyte-colony stimulating factor (G-CSF) + granulocyte macrophage-colony stimulating factor (GM-CSF)
  Interventions: Drug: Etoposide; Drug: G-CSF; Drug: GM-CSF; Drug: Isophosphamide; Drug: Rituximab; Procedure: Apheresis
- Rituximab + Ifosfamide + Etoposide + 1 Growth Factor (Experimental): Growth Factor = granulocyte-colony stimulating factor (G-CSF)
  Interventions: Drug: Etoposide; Drug: G-CSF; Drug: Isophosphamide; Drug: Rituximab; Procedure: Apheresis

INTERVENTIONS:
Drug: Etoposide — 150 mg/m^2 given intravenously over 2 hours every 12 hours x 6 doses.
  Other Names: Vepesid
Drug: G-CSF — Starting dose on day +6 at 6 mcg/kg injection every 12 hours until completion of apheresis.
  Other Names: Filgrastim; Neupogen
Drug: GM-CSF — 250 mcg/m^2 injection given every evening till the completion of apheresis.
  Other Names: Sargramostim; Leukine
  Arms: Rituximab + Ifosfamide + Etoposide + 2 Growth Factors
Drug: Isophosphamide — 10 g/m^2 given intravenously continuous infusion over 72 hours.
  Other Names: ifosfamide; Ifex
Drug: Rituximab — Days +1 (375 mg/m^2) and +8 (1000 mg/m^2) given intravenously.
  Other Names: Rituxan
Procedure: Apheresis — Peripheral blood stem cell collection.

SUMMARY:
Primary Objectives:

1. To determine the efficacy of in vivo purging achieved by rituximab in the two groups.
2. To determine the number of apheresis procedures, total stem cell yield/kg patient body weight and the toxicity profile in the two groups.

Secondary Objectives:

1. To determine the degree of expression of various adhesion molecules in the 2 groups and correlate with time to engraftment of neutrophils, platelets, and red blood cells, efficacy of stem cell mobilization and purging.
2. To determine the incidence of disease progression/relapse at 12 months in the two groups.

DETAILED DESCRIPTION:
Granulocyte-colony stimulating factor (G-CSF) and granulocyte macrophage-colony stimulating factor (GM-CSF) are synthetic (man-made) versions of substances naturally produced in your body. These substances, called colony stimulating factors, help the bone marrow to make new white blood cells. When certain cancer medicines fight your cancer cells, they also affect those white blood cells that fight infection. To help decrease the risk of infections when these cancer medicines are used, colony stimulating factors may be given. Colony stimulating factors are also used to help the bone marrow recover after bone marrow transplantation and stem cell transplantation. They are also used to increase the stem cell count in the blood so that adequate number of stem cells can be collected for purposes of transplantation.

Before the study begins, you will have a complete physical exam and have blood (around 1-2 tablespoons) and urine collected for routine tests. You will have x-rays and CT scans to check on the status of the disease. A sample of bone marrow will be collected for tests. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. Your heart and lung function will be evaluated. You will have an electrocardiogram (ECG - a test that measures the electrical activity of the heart) and either a echocardiogram or a multigated acquisition scan (MUGA) (these are tests that measure heart functions). You will also have lung function tests. Women who are able to have children must have a negative blood or urine pregnancy test.

You will have a plastic tube (central venous catheter - CVL) inserted under your collarbone. The CVL will be left in place for the duration of the treatment. The catheter will be used to deliver most of the drugs and for the collection and transfusion of the stem cells. When possible, all drugs that need to be given by vein will be given using the catheter.

All treatment will be given at M. D. Anderson. First, you will be given chemotherapy to increase the number of stem cells in your blood stream. This chemotherapy will include the drugs ifosfamide, etoposide, and rituximab. You will receive a higher dose of rituximab than is standard of care. The drug ifosfamide will be started on Day 2 and will be given as a continuous injection into a vein over 72 hours. The drug etoposide will also be started on Day 2 and will be given by vein over 2 hours every 12 hours. Rituximab will be given by vein over 4-6 hours on Days 1 and 8. To help decrease the risk of developing side effects caused by the chemotherapy, you will be given fluids by vein and a drug called mesna. Mesna will be given by vein over 24 hours after treatment with ifosfamide is finished. You will have to stay in the hospital for 4-6 days for this part of the treatment.

You will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in one group will receive G-CSF and GM-CSF. Participants in the other group will receive G-CSF alone.

After completion of chemotherapy, you will get GM-CSF and G-CSF or just G-CSF injections (given under the skin) twice a day. These drugs are given to help increase the number of white blood cells and will continue to be given until an adequate number of stem cells have been collected. During this time, you will have blood collected for tests (around 1 tablespoon) at least 3 times a week. If your doctor feels it is necessary, you may have blood collected more often.

Blood stem cells will be collected when your blood counts have returned to normal (about 10-16 days after the chemotherapy). The process of stem cell collection takes about 4 hours. It may take 1-6 sessions to collect the number of stem cells needed for the transplant. The process of stem cell collection is called apheresis. A machine is attached to the catheter under the collar bone and blood is withdrawn. The blood then flows through the machine, which removes stem cells from the blood. The blood is then returned back to you through the catheter. The stem cells are then frozen and stored. These stem cells will be given back to you after the next phase of treatment to help your blood counts recover after high dose chemotherapy. After enough stem cells have been collected, you will be admitted to the hospital for high dose chemotherapy.

You will have check-up visits at various times over the next year as part of your standard evaluation after transplantation to check on the status of the disease.

This is an investigational study. All of the drugs used in this study are FDA approved and are commercially available. Up to 100 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed CD20 positive B-cell non-Hodgkin's lymphoma who are candidates for autologous stem cell transplantation.
2. Age up to 70 years
3. Platelet count > 100,000 mm3, independent of transfusion support
4. Absolute neutrophil count (ANC) > 1500/mm3
5. Zubrod performance status of 2 or less.
6. Negative pregnancy test in women
7. Less than 10% marrow involvement with lymphoma within 4 weeks of study enrollment as defined by bilateral bone marrow aspirations and biopsies.
8. Should be seronegative for HIV, HTLV, hepatitis B surface antigen, hepatitis C antibody.

Exclusion Criteria:

1. Clinical or radiographic evidence of active CNS disease
2. Severe concomitant medical or psychiatric illness
3. Lactating or breast feeding females
4. Less than 3 weeks from the first day of last chemotherapy
5. Prior myeloablative therapy with autologous bone marrow or stem cell rescue
6. Serum bilirubin > 1.5 X ULN, Serum transaminases > 2XULN.
7. Serum creatinine >1.6 mg/dl
8. History of pelvic radiation
9. Patients should not have received more than 3 prior chemotherapy regimens (excluding radiation)
10. Patients should not have received more than 6 cycles of fludarabine therapy

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chitra M. Hosing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hosing C, Munsell MF, Reuben JM, Popat U, Lee BN, Gao H, Korbling M, Shpall EJ, Kebriaei P, Alousi A, De Lima M, McMannis J, Qazilbash M, Anderlini P, Giralt S, Champlin RE, Khouri I. A randomized study comparing chemotherapy followed by G-CSF alone or in combination with GM-CSF for mobilization of peripheral blood stem cells in patients with non-Hodgkin's lymphomas. J Blood Med. 2010;1:49-55. doi: 10.2147/JBM.S9846. Epub 2010 Apr 14. PMID 22282683
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 02/12/2004 through 07/13/2007. All participants recruited at U.T. M.D. Anderson Cancer Center and participating institutions.
Period: Overall Study
Arm/Group | Rituximab + Ifosfamide + Etoposide + 2 Growth Factors | Rituximab + Ifosfamide + Etoposide + 1 Growth Factor
Started | 41 | 43
Completed | 41 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab + Ifosfamide + Etoposide + 2 Growth Factors | Rituximab + Ifosfamide + Etoposide + 1 Growth Factor | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Customized [Number; unit: participants]
  Between 20 and 39 years | 3 | 4 | 7.0
  Between 40 and 59 years | 26 | 29 | 55.0
  Between 60 and 79 years | 12 | 10 | 22.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31.0
  Male | 24 | 29 | 53.0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 43 | 84.0

OUTCOME MEASURES:

1. Primary Outcome: CD34+ Cells/kg in Blood Stem Cells
Description: After blood counts return to normal, stem cell collection (takes approximately 4 hours) up to 6 sessions.
Time Frame: The process of stem cell collections take about 4 hours, 1-6 sessions may be needed.
Measure: Median (Full Range); unit: CD34+ cells/kg
Arm/Group | Rituximab + Ifosfamide + Etoposide + 2 Growth Factors | Rituximab + Ifosfamide + Etoposide + 1 Growth Factor
Number analyzed (Participants) | 41 | 43
CD34+ cells/kg | 7.5 [0.7 to 73] | 10.34 [0.14 to 59]

ADVERSE EVENTS:
Time Frame: 4 years and 3 months
Arm/Group | Rituximab + Ifosfamide + Etoposide + 2 Growth Factors | Rituximab + Ifosfamide + Etoposide + 1 Growth Factor
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43
Other Adverse Events (participants affected / at risk) | 10/41 | 10/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Ifosfamide + Etoposide + 2 Growth Factors (N=41) | Rituximab + Ifosfamide + Etoposide + 1 Growth Factor (N=43)
CYTOKINE RELEASE SYNDROME (Blood and lymphatic system disorders) | 2 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 7 | 6
NAUSEA/VOMITING (Gastrointestinal disorders) | 0 | 2
ANEMIA (Blood and lymphatic system disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes